CLINICAL TRIAL: NCT05248815
Title: Knee Extensor Muscle Strength and Physical Function Before and After Total Knee Replacement
Brief Title: Muscle Strength and Total Knee Replacement
Status: Completed | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: Muscle strength and TKP
Record Dates: First submitted 2022-02-09; First posted 2022-02-21 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2024-11

CONDITIONS: Arthropathy of Knee; Osteo Arthritis Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Patients scheduled for total knee replacement.

SUMMARY:
Purposes: To compare knee extensor muscle strength, physical function and self-reported function before and after total knee replacement with healthy age-matched controls. To describe changes in knee extensor muscle strength up to one year after surgery. To study the relationship between changes in knee extensor muscle strength and changes in physical function, self-reported function and physical activity level and the relationship between changes in knee extensor muscle strength and satisfaction.

Methods: A prospective observational study and comparison with controls. 50-55 individuals aged 65 or older, scheduled for total knee arthroplasty will be recruited to the study group. Measurement of study group 0-2 weeks before surgery and 3, 6 and 12 months following surgery. Comparison with 50-55 healthy age-matched controls.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for total knee replacement on the basis of osteoarthritis of the knee
* Expected rehabilitation in a primary care setting

Exclusion Criteria:

* Difficulties reading or speaking Swedish
* Revision surgery
* Rehabilitation in other settings than primary care

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Participants will be recruited from Alingsås Hospital which is located in the Västra Götaland Region of Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Changes in knee extensor muscle strength of the affected side from before surgery to one year after surgery | Comparison of data before surgery (0-2 weeks) with data 3, 6 and 12 months after surgery
  Maximum voluntary isometric contraction measured using the "make" method with hand-held dynamometry fixated in a knee extension strength training apparatus. Force measurement in Newtons.
Comparison of knee extensor muscle strength of the affected side before surgery with controls | Comparison of data before surgery (0-2 weeks) with data data from the control group
  Maximum voluntary isometric contraction measured using the "make" method with hand-held dynamometry fixated in a knee extension strength training apparatus. Force measurement in Newtons.
Comparison of knee extensor muscle strength of the affected side one year after surgery with controls | Comparison of data one year after surgery with data data from the control group
  Maximum voluntary isometric contraction measured using the "make" method with hand-held dynamometry fixated in a knee extension strength training apparatus. Force measurement in Newtons.
Comparison of knee extensor muscle strength of the affected side with the unaffected side | Before surgery (0-2 weeks). 3, 6 and 12 months after surgery.
  Maximum voluntary isometric contraction measured using the "make" method with hand-held dynamometry fixated in a knee extension strength training apparatus. Force measurement in Newtons.

SECONDARY OUTCOMES:
Comparison of 30 s chair stand test between study group and control group | Comparison of data for the study group from before surgery (0-2 weeks) and 12 months after surgery with data from the control group
  30 s chair stand test measures the number of complete stands the test person is able to perform within 30 s.
Comparison of Knee injury and Osteoarthritis Outcome Score between study group and control group | Comparison of data for the study group from before surgery (0-2 weeks) and 12 months after surgery with data from the control group
  Knee Injury and Osteoarthritis Outcome Score is a self-reported outcome questionnaire that measures 5 sub-scales: pain, other symptoms, function in daily living, function in sport and recreation and knee-related quality of life.
Comparison of 6-min walk test between study group and control group | Comparison of data for the study group from before surgery (0-2 weeks) and 12 months after surgery with data from the control group
Correlation between changes in knee extensor muscle strength of the affected side before and after surgery with changes in 30 s chair stand test, Knee injury and Osteoarthritis Outcome Score, 6-min walk test and physical activity level | Before surgery (0-2 weeks) and 12 months after surgery
  Physical activity level will be measured as activity minutes using a questionnaire.
Correlation between changes in knee extensor muscle strength of the affected side before and after surgery with overall satisfaction one year after surgery | Changes in muscle strength from before surgery (0-2 weeks) and 12 months after surgery, satisfaction 12 months after surgery
  Satisfaction will be measured using a 4-point likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Anette Larsson, PhD, Principal Investigator — Närhälsan Rehabilitering
Locations (3):
- Sweden (3):
  - Närhälsan Sörhaga Rehabmottagning, Alingsås
  - Närhälsan Herrljunga Rehabmottagning, Herrljunga
  - Närhälsan Lerum Rehabmottagning, Lerum

IPD SHARING:
Plan to Share IPD: No